CLINICAL TRIAL: NCT04726267
Title: Incidence of Complete Posterior Vitreous Detachment After Trabeculectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, KKU Eye Center, Department of Ophthalmology, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HE631456
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Posterior Vitreous Detachment
Keywords: posterior vitreous detachment; trabeculectomy; vitreomacular interface
MeSH Terms: conditions — Vitreous Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glaucoma patients who was scheduled for trabeculectomy (Other): Wide-field OCT was performed 1-2 weeks before the trabeculectomy. The OCT was done postoperatively at 1 month, 3 months, 6 months and 12 months after surgery.
  Interventions: Device: Wide-field optical coherence tomography

INTERVENTIONS:
Device: Wide-field optical coherence tomography — Merged 4 images of wide-field optical coherence tomography, 2 images of vertical scan and 2 images of horizontal scan.

SUMMARY:
Intraocular surgery could induce vitreous degeneration and posterior vitreous detachment (PVD). Vitreomacular interface (VMI) abnormalities usually are caused by abnormal PVD, vitreoschisis and partial-thickness PVD. Furthermore, the PVD could induce the peripheral break. The incidence of peripheral break and epimacular membrane (EMM) after pneumatic retinopexy were 11.7% and 4-11%, respectively. Although multiple intravitreal anti-vascular endothelial growth factor (anti-VEGF) injections induced PVD of 5.6%, but peripheral break was reported as only 0.67%.

The most common intraocular surgery is cataract surgery. From the literature review, many methods were used to detect the PVD after phacoemulsification. The former studies used indirect ophthalmoscopy and ocular ultrasound for diagnosis of PVD. The later studies used the optical coherence tomography (OCT) for PVD detection. The OCT device had higher effectiveness in evaluation of the posterior segment, then it can detect post-phacoemulsification PVD more and early than previous studies. Ivastinovic et al demonstrated 59.2% of patients had PVD at 1 month after phacoemulsification, and increased up to 71.4% at 3 months. The incidence of rhegmatogenous retinal detachment (RRD) after phacoemulsification is gradually increased with time. The accumulative risk of RRD was increased from 0.27% at 1 year to 1.27% at 20 years after phacoemulsification.

DETAILED DESCRIPTION:
Trabeculectomy is one of the intraocular surgery. Although the volume of intraocular fluid use during the trabeculectomy was much less than used during phacoemulsification, trabeculectomy also could induce the PVD and it's sequelae such as VMI abnormalities. Because the baseline visual acuity of glaucoma patients who were indicated for trabeculectomy usually quite poor, so the sequelae of PVD can cause more visual loss. The incidence of PVD after trabeculectomy has never been published before and nowadays no standard guideline for retinal examination or screening after surgery. Furthermore, Tsukahara et al introduced wide-field OCT-based PVD classification. The new OCT device with higher technology will be useful in PVD detection.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or primary angle closure glaucoma
* Age 18-65 years
* Could be taken the wide-field OCT images
* Written informed consent

Exclusion Criteria:

* History of intraocular inflammation or infection
* History of ocular trauma or head trauma
* History of intraocular surgery such as intravitreal drug injection and cataract surgery
* History of vitreoretinal diseases such as diabetic retinopathy, retinal vascular occlusion and age-related macular degeneration
* History of laser treatment including laser capsulotomy and retinal photocoagulation
* High myopia; spherical equivalence >4 diopters
* Complete PVD was detected before the enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of PVD | 12 months
  complete PVD

SECONDARY OUTCOMES:
The incidence of VMI abnormalities | 12 months
  Vitreomacular traction, Epimacular membrane, Peripheral retinal break

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No